CLINICAL TRIAL: NCT00609388
Title: Evaluation of Tacrolimus (Prograf®) Intraportal Infusion During the Implantation and the Protective Effect on Ischemia-reperfusion Injury in Orthotopic Liver Transplant Recipients - Single Center Study
Brief Title: Tacrolimus During the Implantation and the Effect on Ischemia-reperfusion Injury in Liver Transplantation
Acronym: TAC-Infusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Martin Bodingbauer, Medical University of Vienna / Dep. of Transplantation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TX 001/07
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2007-12

CONDITIONS: Ischemia Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Tacrolimus; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Group A receives an intraportal Tacrolimus-infusion, ATG Induction, Tacrolimus and Steroids.
  Interventions: Drug: Tacrolimus
- B (Placebo Comparator): Group B receives a placebo-Saline solution (0.9%)-Infusion, ATG induction, Tacrolimus and Steroids.
  Interventions: Other: Saline solution 0.9% (250mL)

INTERVENTIONS:
Drug: Tacrolimus — Immunosuppression, intraoperative intraportal infusion of 1ml Tacrolimus with a concentration of 20 ug/mL
  Other Names: PROGRAF
  Arms: A
Other: Saline solution 0.9% (250mL) — intraoperative intraportal infusion of Saline solution 0.9% (250mL)
  Arms: B

SUMMARY:
The evaluation of the efficacy of an intraportal infusion with Tacrolimus, at the time of liver graft implantation, compared to a control group without immunosuppressive intraportal infusion (Placebo: Saline solution 0.9%) with respect to the initial liver function measured by the parameters of the liver function (LFP): AST (U/L), ALT (U/L), total Bilirubin (mg/dL) and the coagulation factors: NT (%), PTT (s), INR.

ELIGIBILITY:
Inclusion Criteria:

* Multi organ transplantation or retransplantation
* ABO incompatible donor organ recipients- Patients, who are listed on the liver transplant-waiting list at the Vienna General Hospital and who fulfill the clinical requirements (local allocation)
* Written informed consent
* Age > 18
* First transplantation

Exclusion Criteria:

* Fulminant failure of the liver
* Liver-Living donor recipients
* pregnant or nursing women
* Allergy/Intolerance to antimetabolites, HCO-60, EL Cremophor or similar compounds,Steroids or macrolide antibiotics
* HIV-positive donors or recipients
* Participants of another clinical study
* Patient has any form of substance abuse, psychiatric disorder or condition, which, in the opinion of the investigator, may invalidate communication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
initial liver function measured by the parameters of the liver function (LFP): AST (U/L), ALT (U/L), total Bilirubin (mg/dL) and the coagulation factors: NT (%), PTT(s),INR. | Day 1,2,3; Weeks 6 and 12 post OLT

SECONDARY OUTCOMES:
Serum parameters: TNF alpha, IL1, IL6 | within the first 3 month
Histopathology (before and after reperfusion) | within the first 3 month
Frequency of rejection episodes | within the first 3 month
Graft function (Serum) und graft survival at 3 months post Tx | within the first 3 month
Patient survival at 3 months post Tx | within the first 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bodingbauer, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- General Hospital Vienna, Vienna, Austria

REFERENCES:
- [Result] St Peter SD, Post DJ, Rodriguez-Davalos MI, Douglas DD, Moss AA, Mulligan DC. Tacrolimus as a liver flush solution to ameliorate the effects of ischemia/reperfusion injury following liver transplantation. Liver Transpl. 2003 Feb;9(2):144-9. doi: 10.1053/jlts.2003.50018. PMID 12548508
- [Derived] Kristo I, Wilflingseder J, Kainz A, Marschalek J, Wekerle T, Muhlbacher F, Oberbauer R, Bodingbauer M. Effect of intraportal infusion of tacrolimus on ischaemic reperfusion injury in orthotopic liver transplantation: a randomized controlled trial. Transpl Int. 2011 Sep;24(9):912-9. doi: 10.1111/j.1432-2277.2011.01284.x. Epub 2011 Jun 14. PMID 21672049